CLINICAL TRIAL: NCT02644317
Title: Chung Shan Medical University Hospital Institutional Review Board
Brief Title: The Balance Influence of Shoe Inserts on Motor Development Delayed Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, GCRC, Director, Clinical Research, Chung Shan Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CS15103
Record Dates: First submitted 2015-11-30; First posted 2015-12-31 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Development Delay
Keywords: Motor development delay; balance; flatfoot; shoe insert
MeSH Terms: conditions — Learning Disabilities; Psychomotor Disorders; Flatfoot

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- with modified shoe inserts (Experimental): wear the modified shoe inserts and shoes for balance test.
  Interventions: Device: Modified shoe inserts
- without modified shoe inserts (No Intervention): only wear the shoes for balance test.

INTERVENTIONS:
Device: Modified shoe inserts — For experimental arm: wear modified shoe inserts and shoes for balance test.
  Arms: with modified shoe inserts

SUMMARY:
Flatfoot, one of the most common foot problems experienced by preschool-aged children, characterized by the collapse of the foot's medial longitudinal arch. Children with motor developmental delay often have flatfoot, according to clinical observation, and research indicates that preschool age is the main stage of the medial longitudinal arch development period. There flatfoot symptoms due to poor arch shock effect, poor walking endurance, likely to cause gait problems while growing up. The lack of a stable foot structure to support and maintain posture may lead to delayed motor development. Early training intervention and help to balance stability is the main rehabilitation goal for motor developmental delayed children. With understanding of the foot development of motor development delayed children, proper intervention can be provided to improve the movement and stability of the lower limbs. The possible deformation of the foot structure and resultant pain in the future can also be prevented.

DETAILED DESCRIPTION:
The investigators designed a prospective cohort study to long-time follow up of preschool aged children with delayed motor development and to establish standard data, including the foot shape, footprint and balance development. The investigators also discuss the influence of the shoe insert with balance and flatfoot correction. Flatfoot leads to poor gross motor balance and the balance improvement after flatfoot correction has never been studied. The investigators findings should provide direct evidence as a reference for clinical workers.

ELIGIBILITY:
Inclusion Criteria:

* preschool aged children with delayed motor development

Exclusion Criteria:

1. lower limb injury case in six months.
2. other neurological history such as cerebral palsy, traumatic brain injury, spina bifida to cause of developmental delay.
3. have been or are receiving insoles correction or treatment.
4. can not be completed with the instruction by foot measurement and balance measurement.

Ages: 36 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The balance change of Movement ABC-2 scales | baseline/immediately/12 weeks/1 year/2 year
  balance subscore of Movement ABC-2 scales

SECONDARY OUTCOMES:
The change of foot print parameters | baseline/12 weeks/1 year/2 year
  foot-print parameters(using CSI scales)

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Chung Chen, Ph.D., Principal Investigator — School of Physical Therapy, Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan